CLINICAL TRIAL: NCT01250431
Title: Gene Expression Correlates of PTSD Symptom Change After EFT (Emotional Freedom Techniques): A Randomized Controlled Trial
Brief Title: Gene Expression Correlates of Post-Traumatic Stress Disorder (PTSD) Symptom Change After EFT (Emotional Freedom Techniques)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soul Medicine Institute (Other)
Responsible Party: Principal Investigator, Dawson Church, Principal Investigator, Soul Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SMI-YOUNT-11/24/10
Record Dates: First submitted 2010-11-24; First posted 2010-11-30 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFT (Emotional Freedom Techniques) (Experimental): 10 sessions of EFT.
  Interventions: Behavioral: EFT (Emotional Freedom Techniques)
- Wait List (No Intervention): 10 week wait period.

INTERVENTIONS:
Behavioral: EFT (Emotional Freedom Techniques) — 10 EFT sessions
  Arms: EFT (Emotional Freedom Techniques)

SUMMARY:
The purpose of the study is to measure the change in psychological symptoms and gene expression in war veterans after a series of 10 EFT coaching sessions. Outcome studies have shown statistically significant reductions in depression, anxiety, and PTSD in veterans after EFT, and this study extends earlier research using biological sampling. EFT is a form of Energy Psychology (EP) that is sometimes referred to as "emotional acupuncture." It involves self-stimulation of 14 acupuncture points at the end of meridians with the fingertips, while recalling an emotional event such as a combat trauma. It is typically effective in 6 to 15 coaching sessions, making it an efficient clinical technique for reducing affect.

DETAILED DESCRIPTION:
There is peer-reviewed published experimental evidence showing that (a) acupuncture reduces the fear response in the brain, especially the limbic system, and most particularly the amygdala; that (b) tapping or rubbing acupuncture points (acupressure) can be as effective as needling them; that (c) EFTs use of such acupressure is efficacious in reducing anxiety, PTSD and other mood disorders; that (d) EFT reliably reduces emotional intensity associated with traumatic memories, is safe and low-risk; that (e) all EP studies that included a long-term follow-up show that patient gains are maintained over time; that (f) the psychological questionnaires used in this study are validated and safe; and that for all these reasons (g) EP is a treatment of choice among therapists when dealing with the traumatic memories of clients. This study extends these findings by noting changes in gene expression associated with the remission of PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Military Service
* The ability to follow instructions, complete written forms, understand English, and provide informed consent. Subjects are required to be literate and understand English.
* Remaining under the care of a primary care provider such as a VA hospital throughout the entire period of the study
* Between 18 and 80 years old. No children will be research subjects in this study.

Exclusion Criteria:

* A current or past physical or psychiatric disorder that would preclude their being able to respond to the psychosocial measures adequately, or to give blood safely (i.e. cognitive dysfunction, psychosis, or any blood or bleeding disorder)
* Regularly work a night or graveyard shift (to avoid effects of alterations in circadian rhythm)
* Inability to come into the San Francisco laboratory for an afternoon for testing
* Immunomodulatory disorders (e.g. AIDS, rheumatoid arthritis, multiple sclerosis, lupus) or cancer history
* Aggressive chronic periodontitis
* Antibiotics within the last 3 months prior to the recruitment date
* A score of more than 4 on questions 34 and 35 of the SA-45:

Having urges to beat, injure, or harm someone Having urges to break or smash things

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
QRT-PCR Assessment of Gene Expression Associated with Psychological Symptoms of Traumatic Stress | Pre-intervention and Post-intervention
  For the experimental group, the first data point is immediately before the first EFT (Emotional Freedom Techniques) session. The second data point is immediately after the last of 10 weekly sessions. The control group is assessed at intake, and after 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dawson Church, PhD, Principal Investigator — Soul Medicine Institute; Garret Yount, PhD, Principal Investigator — Soul Medicine Institute
Locations (1):
- Soul Medicine Institute, Santa Rosa, California, United States

REFERENCES:
- [Result] Church D, Yount G, Rachlin K, Fox L, Nelms J. Epigenetic Effects of PTSD Remediation in Veterans Using Clinical Emotional Freedom Techniques: A Randomized Controlled Pilot Study. Am J Health Promot. 2018 Jan;32(1):112-122. doi: 10.1177/0890117116661154. Epub 2016 Aug 12. PMID 27520015